CLINICAL TRIAL: NCT01698229
Title: Collection of Cerebrospinal Fluid in Healthy Children
Status: Terminated | Type: Observational
Why Stopped: Study interest shifted
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1111012024
Record Dates: First submitted 2012-08-15; First posted 2012-10-02 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Late Infantile Neuronal Ceroid Lipofuscinosis; Batten Disease
Keywords: Cerebrospinal fluid; Lumbar puncture; Spinal tap; Late infantile neuronal ceroid lipofuscinosis; Batten disease
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 5 mL of cerebrospinal fluid (CSF) will be collected in this study at one time point.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Study cohort is comprised of healthy children, ages 2yrs - 8yrs, who are already undergoing a lumbar puncture procedure at New York Presbyterian Hospital for clinical or diagnostic purposes.
  Interventions: Other: Group 1

INTERVENTIONS:
Other: Group 1 — Collecting a small amount of cerebrospinal fluid (5 mL) from healthy children, ages 2 yrs - 8 yrs, who are already undergoing a lumbar puncture procedure at New York Presbyterian Hospital for clinical or diagnostic purposes.

SUMMARY:
The purpose of this study is to obtain cerebrospinal fluid from healthy children already undergoing a lumbar puncture procedure at New York Presbyterian Hospital, to act as healthy controls when compared to children with late infantile neuronal ceroid lipofuscinosis (LINCL), a fatal neurodegenerative disease.

DETAILED DESCRIPTION:
obtain cerebrospinal fluid from healthy children already undergoing a lumbar puncture procedure at New York Presbyterian Hospital, to act as healthy controls when compared to children with late infantile neuronal ceroid lipofuscinosis (LINCL), a fatal neurodegenerative disease.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ages 2 yrs to 8 yrs
* Children already undergoing a lumbar puncture procedure for clinical or diagnostic purposes

Exclusion Criteria:

* Presence of any significant neurological diseases, as judged by the co-investigators
* Presence of any significant medical conditions including cancer

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects will be healthy controls (children ages 2 years to 8 years) undergoing a lumbar puncture at New York Presbyterian Hospital, for clinical care purposes. They will be inpatients and outpatients.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cerebrospinal fluid (CSF) | 1 time point (once)
  The primary study endpoint is the metabolic profiling of 32 samples of cerebrospinal fluid from healthy subjects, in comparison to 32 samples of CSF from children with LINCL, to determine whether there are biomarkers found in the cerebrospinal fluid that are associated with LINCL.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College / New York Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No